CLINICAL TRIAL: NCT06897748
Title: A Phase II, Multicentre, Randomised, Double-blind, Parallel-group, Placebo-controlled Study to Evaluate the Efficacy and Safety of Tozorakimab in Participants With Symptomatic Chronic Obstructive Pulmonary Disease (COPD) With a History of COPD Exacerbations and Elevated Eosinophils (COMETA)
Brief Title: A Study to Investigate Efficacy and Safety of Tozorakimab Injections Compared With Placebo in Adult Participants With Symptomatic Chronic Obstructive Pulmonary Disease (COPD) With a History of COPD Exacerbations and Elevated Eosinophils
Acronym: COMETA
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AZ-RU-00008
Record Dates: First submitted 2025-03-18; First posted 2025-03-27 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Chronic Obstructive Pulmonary Disease; COPD; tozorakimab; MEDI3506; ICS; LABA/LAMA; Biologic; Biologic Treatment
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tozorakimab (Experimental): Dosing subcutaneously tozorakimab
  Interventions: Drug: Tozorakimab
- Placebo (Placebo Comparator): Dosing subcutaneously with equivalent volume to tozorakimab
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Placebo administered subcutaneously, equivalent volume to tozorakimab throughout the study
  Arms: Placebo
Drug: Tozorakimab — Administered subcutaneously tozorakimab and placebo throughout the study
  Arms: Tozorakimab

SUMMARY:
The purpose of this study is to investigate lung function parameters, composite endpoint for exacerbations in chronic obstructive pulmonary disease (COPDCompEx), symptoms and to provide safety information after tozorakimab or placebo administrations in participants with symptomatic chronic obstructive pulmonary disease (COPD) with history of exacerbations and high blood eosinophil counts.

Study details include the following:

* The maximum duration of the screening/run-in period is 5 weeks. An additional unscheduled visit may be performed prior to randomization to repeat safety assessments as deemed necessary by the investigator.
* Eligible patients will enter 12-week treatment (intervention) period with site visits and investigational product (IP) administration every 2 weeks.
* Participants who complete a treatment period, and have not been prematurely discontinued from IP, will enter a 10-week post-intervention follow-up period.
* The study duration will be 27 weeks at maximum for each participant.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be ≥ 40 years of age and capable of giving signed informed consent.
2. Documented diagnosis of COPD for at least one year prior to enrolment.
3. Post-BD FEV1/FVC < 0.70 and post-BD FEV1 >20% and < 80% of predicted normal value.
4. Documented history of ≥ 2 moderate or ≥ 1 severe COPD exacerbations within 12 months prior to enrolment.
5. Documented optimised inhaled dual or triple therapy for at least 3 months prior to enrolment.
6. Smoking history of ≥ 10 pack-years.
7. CAT total score ≥ 10, with each of the phlegm (sputum) and cough items with a score ≥ 2.
8. All participants must have eosinophil blood count ≥ 150 cells/µL.

Exclusion Criteria:

1. Clinically important pulmonary disease other than COPD.
2. Radiological findings suggestive of a respiratory disease other than COPD that is significantly contributing to the participant's respiratory symptoms. Radiological findings of pulmonary nodules suspicious for lung cancer, as per applicable guidances, without appropriate follow up prior to randomisation. Radiological findings suggestive of acute infection.
3. Current diagnosis of asthma, prior history of asthma, or asthma-COPD overlap. Childhood history of asthma is allowed and defined as asthma diagnosed and resolved before the age of 18.
4. Any unstable disorder, including, but not limited to, cardiovascular, gastrointestinal, hepatic, renal, neurological, musculoskeletal, infectious, endocrine, metabolic, haematological, psychiatric disorder, major physical and/or cognitive impairment that could affect safety, study findings or participants ability to complete the study.
5. COPD exacerbation, within 2 weeks prior to randomization, that was treated with systemic corticosteroids and/or antibiotics, and/or led to hospitalization.
6. Active significant infection within the 4 weeks prior to randomization, pneumonia within 6 weeks prior to randomization, or medical condition that predisposes the participant to infection.
7. Significant COVID-19 illness within the 6 months prior to enrolment.
8. Unstable cardiovascular disorder.
9. Diagnosis of clinically significant cor pulmonale, pulmonary arterial hypertension and/or right ventricular failure.
10. History of active severe inflammatory bowel disease or colitis within one year prior to enrolment, or unexplained diarrhoea within the 4 weeks prior to randomisation.
11. History of known immunodeficiency disorder, including a positive test for HIV-1 or HIV 2.
12. History of positive test or treatment for hepatitis B or hepatitis C (except for cured hepatitis C).
13. Evidence of active liver disease, including jaundice during screening.
14. Malignancy, current or within the past 5 years, except for adequately treated non-invasive basal cell and squamous cell carcinoma of the skin and cervical carcinoma-in-situ treated with apparent success more than one year prior to enrolment. Suspected malignancy or undefined neoplasms.
15. Participants who, in the opinion of the Investigator or qualified designee, have evidence of active TB.
16. History of partial or total lung resection.
17. Scheduled major surgical procedure during the course of the study.
18. Participants that have previously received tozorakimab.
19. Change in smoking status in 12 weeks prior to enrolment or intention to change smoking status between enrolment and end of follow-up.
20. Any clinically significant abnormal findings in physical examination, vital signs, ECG, or laboratory testing during the screening period, which in the opinion of the investigator may put the participant at risk because of their participation in the study, or may influence the results of the study, or the participant's ability to complete the entire duration of the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2025-04-12 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline to Week 12 in Pre-bronchodilator Forced Expiratory Volume in 1 Second (Pre-BD FEV1) as Measured in Clinic | Baseline through Week 12
  The difference in mean change from baseline in FEV1

SECONDARY OUTCOMES:
Annualized rate of composite endpoint for exacerbations in COPD (COPDCompEx) events | From baseline to Week 12
  The rate ratio of COPDCopmEx events
Change from baseline in post-BD FEV1 | From baseline through Week 12
  The difference in mean change from baseline in post-BD FEV1
Change from baseline in pre-BD and post-BD forced vital capacity (FVC) | From baseline through Week 12
  The difference in mean change from baseline in pre-BD and post-BD FVC
FEV1 % reversibility dynamics | From baseline to Week 12
  The difference in mean change from baseline in FEV1 % reversibility
Change from baseline in peak expiratory flow (PEF) measured in clinic and at home | From baseline through Week 12
  The difference in mean change from baseline in PEF
Change from baseline in home FEV1 | From baseline through Week 12
  The difference in mean change from baseline in FEV1
Time to first COPDCompEx event | From baseline to Week 12
  The hazard ratio for COPDCompEx event occurrence
Change from baseline in mean Breathless, cough and sputum scale (BCSS) score | From baseline to Week 12
  The difference in mean change from baseline in BCSS.
  The BCSS, is a 3-item daily Diary that assesses the severity of the 3 symptoms: breathlessness, sputum, and cough; each on a 5-point scale (from 0 to 4). Higher scores for each domain, and thus for total score, indicate more severe symptoms.
Change from baseline in COPD assessment test (CAT) total score | From baseline to Week 12
  The difference in mean change from baseline in CAT.
  The CAT consists of eight questions that ask the participant to rate items relating to symptoms and impact on quality of life (such as normal activity and sleep). Each question is performed on a scale from 0 to 5 with 0 being the best possible health status or least impairment and 5 being the worst health status or greatest impairment.

OTHER OUTCOMES:
Number of patients with adverse events (AEs) | Through study completion, up to 27 weeks
  The measure of interest is frequencies and percentages of participants with reported AEs.

CONTACTS AND LOCATIONS:
Locations (9):
- Russia (9):
  - Research Site, Aramil
  - Research Site, Izhevsk
  - Research Site, Moscow
  - Research Site, Omsk
  - Research Site, Penza
  - Research Site, Perm
  - Research Site, Saint Petersburg
  - Research Site, Saratov
  - Research Site, Ulyanovsk

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at :
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home